CLINICAL TRIAL: NCT03147807
Title: BetaLACTA® Test-guided Early De-escalation of Empirical Carbapenems in Pulmonary, Urinary and Bloodstream Infections Diagnosed in Intensive Care Unit - BLUE¬-CarbA Study
Brief Title: BetaLACTA® Test for Early De-escalation of Empirical Carbapenems in Pulmonary, Urinary and Bloodstream Infections in ICU
Acronym: BLUE-CarbA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 150940; N° IDRCB 2016-A00941-50 (Other: AOM 15470)
Record Dates: First submitted 2017-02-02; First posted 2017-05-10 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Pneumonia; Urinary Tract Infections; Bloodstream Infection
Keywords: Carbapenems de-escalation, rapid diagnostic test,; Carbapenem-antimicrobial de-escalation-rapid diagnostic test
MeSH Terms: conditions — Pneumonia; Urinary Tract Infections; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- betaLACTA® result given to physician (Experimental): In the experimental group, betaLACTA® rapid diagnostic test guided de-escalation result will be given to physician at Day 0 and empirical carbapenems will be de-escalated to Cefepime or Ceftazidime +/- Amikacin since the second dose.
  Interventions: Device: betaLACTA® rapid diagnostic test
- betaLACTA® result NOT given to physician (No Intervention): In the control group, betaLACTA® result will not be given to physician and patients will receive empirical carbapenem during the time required to obtain final results of antibiotic susceptibility test

INTERVENTIONS:
Device: betaLACTA® rapid diagnostic test — Since ≥1 bacteriological sample(s) from ICU patients empirically treated with carbapenems (i.e. respiratory sample such as quantitative tracheobronchial aspirate with available volume ≥1 mL; urinary sample such as single catheter urine specimen; or blood culture) is positive for ≥2 GNB/field on direct examination, empirical carbapenem will be adapted: 1) early, since the second dose, according to the results of the betaLACTA® rapid diagnostic test (BLT) in the intervention arm (i.e. de-escalation to cefepim or to ceftazidim+amikacin in case of negativity, and carbapenem continuation in case of positivity); or 2) after 48-72h according to the results of the antibiotic susceptibility test in the control arm.
  Other Names: betaLACTA® test
  Arms: betaLACTA® result given to physician

SUMMARY:
The emergence and rapid worldwide spread of Extended- Spectrum Beta-Lactamase-producing enterobacteriaceae (ESBLE) both in hospital and community, led physicians, and notably intensivists, to prescribe more carbapenems, particularly in the most fragile patients such as ICU patients. Unfortunately, the increased carbapenem consumption favored the emergence of carbapenem resistance mechanisms. Moreover, several preliminary results suggest that carbapenem could markedly impact the human intestinal microbiota, Thus, reduction of carbapenem exposure is widely desired both by national and international antibiotic plans. Therefore, the use of rapid diagnostic tests evaluating bacterial resistance to reduce inappropriate exposure to carbapenems could be a relevant solution. Due to its good diagnostic performance, the betaLACTA® test could meet these objectives.

Experimental plan :

Randomized, open-labeled non-inferiority clinical trial involving an in vitro diagnostic medical device (close to a phase III study), comparing two parallel groups:

* Experimental group: early carbapenems de-escalation since the second dose, guided by results of the betaLACTA® test performed directly on the bacterial pellet from the microbiological sample positive on direct examination.
* Control group: carbapenems de-escalation guided by definitive results of the antibiotic susceptibility test obtained 48 to 72h after microbiological sampling (reference strategy).

DETAILED DESCRIPTION:
This study is conducted on ICU patients with a suspected pneumonia, primary blood-stream infection (BSI), and/or urinary tract infection (UTI).

The primary objective of the study is to demonstrate that in ICU infections treated empirically by carbapenems and documented with GNB on direct examination of a respiratory, urinary and/or blood sample(s), the early de-escalation guided by the results of the betaLACTA® test is not inferior to the reference strategy de-escalating on antibiotic susceptibility test (AST) results obtained 48-72h after sampling, in terms of mortality at D90 and infection recurrence in ICU.

The secondary objectives are to compare the early de-escalation guided by the betaLACTA® test results to the reference strategy de-escalating on the AST results on:

* The exposure to carbapenems.
* The total use of ICU and hospital resources and the cost-effectiveness.
* The occurrence of other infections.
* The colonization of the digestive tractus of patients with 3rd generation cephalosporins (3rdGC) resistant Gram-negative bacteria (GNB).

In addition, an ancillary study will be performed (only in participating centers from the Ile de France region) to compare :

* The composition of the intestinal microbiota among patients with an early de-escalation guided by the betaLACTA® test results and a standard de-escalation on AST results at 48-72h.
* The evolution of intestinal microbiota of patients after exposure to different beta-lactam antibiotics, from carbapenems or cefepim/ceftazidim during the empirical treatment, to the definitive beta-lactam antibiotic chosen to cure the infection after antibiotic susceptibility test results.
* The outcomes of ICU patients (mortality at D90, occurrence of infection, ICU length of stay, etc.) according to the composition of their intestinal microbiota and to its evolution during antibiotic treatment.

To meet these objectives, 646 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients ≥18 years.
* With a suspected pneumonia (according to CPIS definition), primary blood-stream infection (according to CDC definition), and/or urinary tract infection (according to IDSA Guidelines).
* And presence of ≥2 GNB/field on direct examination of a respiratory sample (quantitative bronchial aspirate with an available volume ≥ 1mL), urinary sample or blood culture.
* Leading to an empirical carbapenem prescription, not administered for more than 6 hours when considering the inclusion of the patient.
* Written informed consent signed by the patient / the trustworthy person / the next-of-kin / close relative, or inclusion in case of emergency and written informed consent will been signed by the patient as soon as possible.
* Patients affiliated to French social security.

Exclusion Criteria:

* Pregnancy.
* Allergy to beta-lactams.
* Patients already treated with ongoing carbapenems for another documented infection, blocking carbapenem de-escalation.
* Patients included in another interventional study.
* Patients in whom a procedure of withdrawing life-sustaining treatment was decided before inclusion.
* Moribund patients.
* Patients with aplasia.
* Patients under tutorship/curatorship or patient deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
mortality at D90 and infection recurrence during the ICU stay | Day 90
  Composite endpoint combining 90-day mortality and percentage of infection recurrence (same GNB on the same site of infection) during the ICU stay (within the limit of 90 days).
  Recurrence will be defined a posteriori by 3 independent experts, blinded of the allocation group of patients in whom a suspected recurrence would have occurred, with predefined criteria.

SECONDARY OUTCOMES:
Exposure to carbapenems | from Day 0, through ICU discharge or until 28 days after inclusion in case of prolonged ICU stay
  * Number of days with carbapenem treatment after inclusion during ICU stay (within the limit of 28 days)
  * Number of carbapenems Defined Daily Doses (DDD) after inclusion during ICU stay (within the limit of 28 days)
  * Number of carbapenem-free and antibiotic free days at day 28 after inclusion
Total use of ICU and hospital resources and cost-effectiveness of early de-escalation compared to standard de-escalation. | from Day 0,throught hospital discharge or until 28 days after inclusion in case of prolonged ICU stay
  * ICU and hospital lengths of stay following randomization;
  * Total cost and incremental cost-effectiveness ratio (cost per additional death/ infection averted).
Occurrence of other infections. | From Day 0 to ICU discharge (within the limit of 90 days).
  Percentage of new infections (same site of infection with other bacteria or other site of infection) during ICU stay (within the limit of 90 days).
Colonization of the digestive tractus of patients with 3rd generation cephalosporins (3rdGC) resistant Gram-negative bacteria | From Day 0, through ICU discharge or until 28 days after inclusion in case of prolonged ICU stay
  New colonization of patients' digestive tractus with 3rdGC-resistant GNB (i.e. ESBL-producing Enterobacteriaceae, Carbapenemase-producing Enterobacteriaceae, high-concentration AmpC cephalosporinase-producing Enterobacteriaceae, multi-resistant non-fermenting GNB, etc.) will be assessed comparing the results of the culture on selective media of rectal swabs performed at inclusion and at D3, at the end of the antibiotic treatment, and at ICU discharge.
  Characterization of acquired 3rdGC-resistant GNB and determination of their resistance mechanism(s) will be performed using standard microbiological processes and molecular biology.
Composition of intestinal microbiota at Day 0 | from D0 to the end of the antimicrobial treatment of the infection leading to inclusion in the study, average 7-10 days
  To compare the composition of intestinal microbiota among patients with an early de-escalation guided by the betaLACTA® test results and a standard de-escalation on antibiogram results at 48-72h.
Composition of intestinal microbiota at day 3 | from D0 to the end of the antimicrobial treatment of the infection leading to inclusion in the study, average 7-10 days
  To compare the evolution of intestinal microbiota of patients after exposure to different betalactam antibiotics, from carbapenems or cefepim/ceftazidim during the empirical treatment, to the definitive beta-lactam antibiotic chosen to cure the infection after antibiotic susceptibility test results.
Composition of intestinal microbiota after antibiotic exposur | from D0 to the end of the antimicrobial treatment of the infection leading to inclusion in the study, average 7-10 days
  To compare the outcomes of ICU patients (mortality at Day 90, occurrence of infection, ICU length of stay, etc.) according to the composition of their intestinal microbiota and to its evolution during antibiotic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Marc GARNIER, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Anesthesiology and Critical Care Medicine Department, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garnier M, Gallah S, Vimont S, Benzerara Y, Labbe V, Constant AL, Siami S, Guerot E, Compain F, Mainardi JL, Montil M, Quesnel C; BLUE-CarbA study group.. Multicentre randomised controlled trial to investigate usefulness of the rapid diagnostic betaLACTA test performed directly on bacterial cell pellets from respiratory, urinary or blood samples for the early de-escalation of carbapenems in septic intensive care unit patients: the BLUE-CarbA protocol. BMJ Open. 2019 Feb 19;9(2):e024561. doi: 10.1136/bmjopen-2018-024561. PMID 30782909